CLINICAL TRIAL: NCT07355881
Title: The Modified SOAR Score as a Predictor of Early Mortality in Hospitalized Patients With Acute Stroke
Brief Title: mSOAR and Early Mortality in Acute Stroke
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Kareman Mohamed Abdelaziz, Principal investigator, Sohag University
Other Study IDs: Soh-Med--25-12-16MS
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Stroke Patients
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — Participants will receive standard of care only. No study-specific intervention is applied.

SUMMARY:
This observational study aims to evaluate the predictive accuracy of the Modified SOAR score for early mortality in patients with acute stroke. Adult patients presenting with acute stroke at Sohag University Hospitals will be included. Data on clinical presentation, medical history, and relevant laboratory investigations will be collected. The study will follow patients during their hospital stay to determine outcomes related to early mortality. The findings will help improve early risk stratification and management of acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute stroke
* Patients admitted to Sohag University Hospitals
* Patients who underwent clinical evaluation
* Patients who provided informed consent

Exclusion Criteria:

* Patients with transient ischemic attack (TIA)
* Patients with orthopedic conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients diagnosed with acute stroke who are admitted to Sohag University Hospitals. Patients must present within 24 hours of symptom onset and provide informed consent. This cohort will include both male and female patients, and patients with complete medical records necessary for calculating the Modified SOAR score.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Early Mortality | 7days
  Assessment of early mortality in patients with acute stroke during the follow-up period.
Early mortality | 7 days
  Assessment of early mortality in patients with acute stroke during the first 7 days of hospital admission. Patients will be monitored from hospital admission until 7 days or until death, whichever occurs first. The Modified SOAR score will be recorded for each patient at admission to evaluate its predictive accuracy for early mortality within this period.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No